CLINICAL TRIAL: NCT00795834
Title: Pilot Study to Assess Effects of Novel Beverages on Established and Novel Risk Markers for Vascular Disease
Brief Title: Effects of a Beverage Rich in Fruit Extracts on Risk Factors Associated With Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Professor Naveed Sattar, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 07/S0704/110; RN08BI013
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: Cardiovascular Disease
Keywords: polyphenolics; flavonols; lipids; endothelial function; vascular risk factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beverage (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Beverage
- High Polyphenol Beverage (Active Comparator)
  Interventions: Dietary Supplement: High polyphenol beverage

INTERVENTIONS:
Dietary Supplement: High polyphenol beverage — Antioxidant capacity umol TE/L(ORAC): 19987 Polyphenolic Content(mcg/ml): 1445 Vitamin C (mg/100ml): 35.35 Calorie Content (Kcal/250ml):40.0
  250ml twice daily for 1 month (56 doses)
  Arms: High Polyphenol Beverage
Dietary Supplement: Placebo Beverage — Antioxidant capacity umol TE/L(ORAC): negligible Polyphenolic Content(mcg/ml): negligible Vitamin C (mg/100ml): 0.00 Calorie Content (Kcal/250ml):40.0
  250ml twice daily for 1 month (56 doses)
  Arms: Beverage

SUMMARY:
The purpose of this study is to assess the effects of a novel beverage rich in polyphenols (compounds present in fruit extracts) on risk factors associated with cardiovascular disease.

DETAILED DESCRIPTION:
This study will assess the potential of a beverage containing plant and fruit extracts rich in polyphenolics to modulate vascular risk.

Novel risk factors for vascular disease will be assessed including non-invasive assessment of vascular function by pulse wave analysis / pulse wave velocity and laser doppler iontophoresis.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 55 years
* BMI > 25

Exclusion Criteria:

* Present smoker or smoked within the last 2 years
* HBA1C > 6.0%
* eGFR<60
* LFT >/= 3 times upper limit of normal
* Hypertension: systolic blood pressure > 160mmHg; diastolic blood pressure > 90mmHg, or on medication for hypertension.
* Chronic disease, likely to be clinically relevant (eg:

cardiorespiratory, rheumatological, cerebrovascular or neoplastic disease)

* Vitamin supplements within the previous 14 days
* Medications which, in the opinion of the investigators, are known to influence vascular function (eg corticosteroids).

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-01 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Vascular Function (measured by Laser Doppler Iontophoresis and Pulse Wave Analysis / Pulse Wave Velocity) | Baseline and post intervention

SECONDARY OUTCOMES:
Established and novel blood markers for vascular disease | baseline and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Sattar, MBChB PhD FRCPath FRCP, Principal Investigator — University of Glasgow
Locations (1):
- British Heart Foundation Glasgow Cardiovascular Research Centre, Glasgow, United Kingdom

REFERENCES:
- [Derived] Mullan A, Delles C, Ferrell W, Mullen W, Edwards CA, McColl JH, Roberts SA, Lean ME, Sattar N. Effects of a beverage rich in (poly)phenols on established and novel risk markers for vascular disease in medically uncomplicated overweight or obese subjects: A four week randomized placebo-controlled trial. Atherosclerosis. 2016 Mar;246:169-76. doi: 10.1016/j.atherosclerosis.2016.01.004. Epub 2016 Jan 6. PMID 26797134